CLINICAL TRIAL: NCT06601335
Title: A Randomized, Controlled, Multicenter Phase 3 Study of AK112 in Combination With AK117 Versus Pembrolizumab as First Line Treatment for a Programmed Cell Death-ligand 1 (PD-L1) Positive Population With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC)
Brief Title: A Phase 3 Study of AK112 Plus AK117 Versus Pembrolizumab in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK117-302
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK117 in combination with AK112 (Experimental)
  Interventions: Drug: AK117 in combination with AK112
- Placebo in combination with Pembrolizumab (Active Comparator)
  Interventions: Drug: Placebo in combination with Pembrolizumab

INTERVENTIONS:
Drug: AK117 in combination with AK112 — Following a predefined dose and date.
  Arms: AK117 in combination with AK112
Drug: Placebo in combination with Pembrolizumab — Following a predefined dose and date.
  Arms: Placebo in combination with Pembrolizumab

SUMMARY:
This is a phase 3 study. All subjects arerecurrent or metastatic head and neck squamous Cell Carcinoma (R/M HNSCC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the efficacy and safety of AK112 combined with AK117 versus pembrolizumab combined with placebo in patients with R/M HNSCC whose tumors have programmed cell death-ligand 1 (PD-L1) positive [Combined Positive Score (CPS) greater than or equal to 1].

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent.
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Have a life expectancy of at least 3 months.
4. Has histologically confirmed diagnosis of R/M HNSCC primarily located in oropharynx, oral cavity, hypopharynx, or larynx, which is considered incurable by local therapies.
5. Participants with oropharyngeal cancer must have results from testing of human papillomavirus HPV status.
6. No prior systemic treatment for R/M HNSCC.
7. At least one measurable noncerebral lesion according to RECIST 1.1.
8. PD-L1 positive (CPS ≥ 1).
9. Has adequate organ function.
10. All subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.
11. Able to to comply with all requirements of study participation (including all study procedures).

Exclusion Criteria:

1. Has squamous cell carcinoma of the primary site, such as nasopharynx, nasal cavity, sinuses, salivary glands, thyroid or parathyroid, skin, or of unknown primary origin.
2. Had other malignant tumors within the 5 years prior to enrollment.
3. Has a significant risk of bleeding assessed by the investigator based on imaging.
4. Radiologically documented evidence of major blood vessel invasion or tumor invading organs or there is a risk of esophagotracheal or esophagopleural fistula, or major blood vessel encasement that the investigator determines will pose a significantly increased risk of bleeding.
5. Has known active central nervous system (CNS) metastases.
6. Has pleural effusion, pericardial effusion, or ascites with clinical symptoms or requiring repeated drainage.
7. Previously received immunotherapy, including immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy, and any other treatments targeting the immune mechanisms of tumors.
8. Previously received radiation therapy for head or neck within 8 weeks prior to enrollment, received palliative radiation therapy for non-head or non-neck within 3 weeks prior to enrollment.
9. Has a history severe bleeding tendency or coagulation dysfunction.
10. Has a history myocarditis, cardiomyopathy, and malignant arrhythmia.
11. Has a history arterial or venous thromboembolism events, transient ischemic attacks, cerebrovascular accidents, hypertensive crises, or hypertensive encephalopathy occurred within 6 months prior to enrollment.
12. Pregnant or lactating female.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 2 years
  OS is the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented disease progression (per RECIST v1.1 criteria) assessed by investigators or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , assessed by investigators based on RECIST v1.1.
Adverse Events (AEs) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Cmax | Up to approximately 2 years
  Maximum plasma concentration of AK112 and AK117 after administration.
Cmin | Up to approximately 2 years
  Minimum plasma concentration of AK112 and AK117 after administration.
Anti-drug antibodies (ADA) | Up to approximately 2 years
  Number of subjects with detectable ADA.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - West China Hospital of Sichuan University, Chengdu, Sichuan